CLINICAL TRIAL: NCT03428113
Title: Measuring Bladder Volumes With Ultrasound and Bladder Scanning in the ICU
Brief Title: Measuring Bladder Volumes Scanning in the ICU
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Lynn Schallom, Director of Research For Patient Care Services at Barnes-Jewish Hospital, Washington University School of Medicine
Other Study IDs: 201704104
Record Dates: First submitted 2018-01-22; First posted 2018-02-09 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Urinary Retention; Acute Kidney Injury
MeSH Terms: conditions — Urinary Retention; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICU patient unable to void for 6 hours: ICU patients unable to void after 6 hours after a indwelling urinary catheter is removed or since time of admission
  Interventions: Other: Bladder Volume Measurement bladder scanner RN; Other: Bladder Volume Measurement Ultrasound APRN; Other: Bladder Volume Measurement bladder scanner APRN; Other: Bladder Volume Measurement Ultrasound MD; Other: Intermittent Straight Catheterization
- renal failure with low urine volume: ICU patients with renal failure, acute kidney injury or acute on chronic with minimal urine output without an indwelling urinary catheter
  Interventions: Other: Bladder Volume Measurement bladder scanner RN; Other: Bladder Volume Measurement Ultrasound APRN; Other: Bladder Volume Measurement bladder scanner APRN; Other: Bladder Volume Measurement Ultrasound MD; Other: Intermittent Straight Catheterization

INTERVENTIONS:
Other: Bladder Volume Measurement bladder scanner RN — Measure Urine Volume with Bladder Scanner by RN
  Other Names: Bladder Scanner
Other: Bladder Volume Measurement Ultrasound APRN — Measure Urine Volume with Point of Care Ultrasound by APRN
  Other Names: Ultrasound APRN
Other: Bladder Volume Measurement bladder scanner APRN — Measure Urine Volume with Bladder Scanner by APRN
  Other Names: Bladder Scanner APRN
Other: Bladder Volume Measurement Ultrasound MD — Measure Urine Volume with Point of Care Ultrasound by MD
  Other Names: Ultrasound MD
Other: Intermittent Straight Catheterization — Measure Urine Volume with Intermittent Straight Catheterization

SUMMARY:
ICU patients are at risk for catheter associated urinary tract infection. Frequently patients can't tell clinicians if they need to void if the catheter is removed. If clinicians know that an accurate volume measurement s of urine volume in the bladder can be obtained when the catheter is removed, catheters could be removed earlier and more frequently and thus possibly avoid an infection. For this study, measures with ultrasound (directly visualizing the bladder to measure), bladder scanner (partially blind measure with placement of scanner over the expected bladder location on the skin) and urine catheterized volume will be obtained. The investigators also want to know if the technology is user dependent. The study will include 2 levels of nurses RN and advanced practice RN (APRN) perform the bladder scanner. An APRN and MD will conduct the ultrasound. Ultrasound is technology primarily used by physicians but APRNs are using the technology technology more frequently. After these 4 measurements, the patient's nurse will perform an intermittent straight catheterization (catheter inserted, urine drained, and catheter removed) as the gold standard comparison.

DETAILED DESCRIPTION:
The purpose of this correlational descriptive study is to compare measured bladder volumes with a bladder scanner (Verathon Prime), 3D ultrasound (Sono-Site II) and straight catheterization in ICU patients with low urine output receiving dialysis and in ICU patients unable to void.

Upon consent of patient or LAR, patient's age, gender and BMI with the assigned study code number will be recorded on enrollment log. Study code number, patient initials and unit will be written on bedside data collection sheet.

Sequence of 4 non-invasive (1-4) measurement will vary from day to day (see below)

1. MD performs bladder ultrasound and records volume on data collection sheet and places in envelope
2. APRN performs bladder scanner and records volume on data collection sheet and places in envelope.
3. APRN performs bladder ultrasound and records volume on data collection sheet and places in envelope
4. Bedside RN performs bladder scanner and records volume on data collection sheet and places in envelope
5. The study team will record the data from the straight catheterization that is performed as part of clinical care.
6. APRN or research nurse will retrieve catheterization urine volume measurement from RN or from chart and record on data collection sheet

Each enrolled patient will have these 4 measurements performed only on one day. Each clinician research team member will record their result on a data collection form with the study number, patient initials, day of week, clinician initials, observation of abdominal fluid, and comment section for any other observations. The clinician research team member will place the completed form for their measurement in an envelope with the study number on the outside while the next clinician is in the room obtaining the next measure.

Data collection is complete after catheter volume is recorded.

ELIGIBILITY:
Inclusion Criteria:

* ICU dialysis patients who have their catheter removed per ICU medical team
* ICU patients without an indwelling urinary catheter and inability to void 6 hours post urinary catheter removal or 6 hours after admission

Exclusion Criteria:

* Pregnant women Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with low urine output due to new acute kidney injury or patients unable to void, secondary to surgical procedure, change in level of consciousness, or neurological alteration
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Intermittent Straight Catheterization Volume Compared to Bladder Scan Measurement Volume | At time of enrollment, one point in time
  Comparison of the two measurements of bladder volume will be analyzed
Intermittent Straight Catheterization Volume Compared to Point of Care Ultrasound Measurement Volume | At time of enrollment, one point in time
  Comparison of the two measurements of bladder volume will be analyzed

SECONDARY OUTCOMES:
Clinician Level Measurements with Bladder Scanner and Point of Care Ultrasound | At time of enrollment, one point in time
  Comparison of the two measurements between clinicians 1. Bladder Scan measurement by bedside RN compared to APRN bladder scan measurement) and 2. APRN Ultrasound compared to MD US will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes-Jewish Hospital at Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No